CLINICAL TRIAL: NCT03383484
Title: Use of Osteopathic Principles for Nonpharmacologic, Therapeutic Interventions in Women With Polycystic Ovary Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diana Speelman, Ph.D. (Other)
Responsible Party: Sponsor-Investigator, Diana Speelman, Ph.D., Principal Investigator, Lake Erie College of Osteopathic Medicine
Organization: Lake Erie College of Osteopathic Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-156; 181627705 (Other Grant/Funding Number: American Osteopathic Association)
Record Dates: First submitted 2017-12-12; First posted 2017-12-26 (Actual); Last update posted 2017-12-26 (Actual); Status verified 2017-12

CONDITIONS: Polycystic Ovary Syndrome
Keywords: polycystic ovary syndrome; hyperandrogenism; nonpharmacological; yoga; osteopathic manipulative medicine
MeSH Terms: conditions — Polycystic Ovary Syndrome; Hyperandrogenism | interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No intervention (No Intervention): No OMT, yoga, acupuncture, or other interventions.
- OMT intervention (Experimental): Weekly OMT for 3 months
  Interventions: Other: OMT
- Yoga intervention (Experimental): Yoga 3 times per week for 3 months
  Interventions: Other: Yoga

INTERVENTIONS:
Other: OMT — Weekly manipulation of Chapman points and rib raising techniques (osteopathic manipulative treatment)
  Arms: OMT intervention
Other: Yoga — Yoga practice 3 times per week for 1 hour each time; hatha yoga poses, asanas, and breathing techniques
  Arms: Yoga intervention

SUMMARY:
The overall goals of this project are to assess the efficacy of non-pharmacological, complementary therapies to improve outcomes in the treatment of women with polycystic ovary syndrome (PCOS). The studies proposed herein are designed to assess the efficacy of osteopathic manipulative medicine (OMM) in the assessment of sympathetic tone in these women, and the effectiveness of non-pharmacologic therapeutic interventions in improving participant metabolic, endocrine, reproductive, and psychological health.

DETAILED DESCRIPTION:
Question 1: Can osteopathic structural assessment identify increased sympathetic tone in women with PCOS? Specific Aim 1: To use palpation of Chapman points and spinal viscerosomatic reflex regions to assess the presence and degree of increased sympathetic tone in women with PCOS.

Chapman points and viscerosomatic reflexes reflect visceral dysfunction and are mediated by the sympathetic nervous system, and can be a very useful clinical diagnostic tool. There is increased sympathetic tone in women with PCOS as well as in obese individuals, as previously determined by physiologic measures. Increased sympathetic tone in the study population will be assessed by osteopathic structural assessment and confirmed by physiologic measures of heart rate, heart rate variability, resting blood pressure, and blood pressure and heart rate recovery following exercise.

Hypothesis: Chapman points will be palpable at regions for the heart, adrenal glands, and ovaries to indicate hyperactivity of the sympathetic nervous system and will correlate with physiologic evidence of increased sympathetic tone.

Hypothesis: Alterations of viscerosomatic reflexes associated with the heart, adrenal glands, and ovaries will reflect hyperactivity of the sympathetic nervous system and will correlate with physiologic evidence of increased sympathetic tone.

Question 2: Can regular, sympathetic nervous system-targeted osteopathic manipulative treatment (OMT) improve endocrine and reproductive parameters, and sympathetic tone, in women with PCOS? Specific Aim 2: To use weekly manipulation of Chapman points and spinal regions associated with viscerosomatic reflexes in women with PCOS for improvement of endocrine and reproductive parameters, and sympathetic tone, after 3 months of treatment.

Chapman points and viscerosomatic reflexes are useful in diagnosis, and may be manipulated to restore somatovisceral health.

Hypothesis: Completion of 3 months of weekly manipulation of Chapman points and viscerosomatic reflexes will improve sympathetic tone (as assessed by both osteopathic structural assessment and physiologic parameters), androgen levels, and menstrual cycle length compared to women with PCOS and no intervention.

Question 3: Can regular yoga improve metabolic, endocrine, reproductive, and psychological parameters in women with PCOS? Specific Aim 3: To use thrice-weekly yoga practice with mindfulness techniques in women with PCOS to improve metabolic, endocrine, reproductive, and psychological parameters after 3 months of intervention.

The benefits of moderate and high-intensity aerobic activity on metabolic and overall health for women with PCOS have been reported, but the effects of low-impact exercise are less studied. Women with PCOS will participate in a yoga class with integrated mindfulness techniques 3 times per week for 3 months.

Hypothesis: Thrice weekly yoga intervention for 3 months will result in an improvement in androgen levels, fasting blood glucose, menstrual cycle length, and patient-reported anxiety, compared to women with PCOS and no intervention.

ELIGIBILITY:
Inclusion Criteria:

* Females between the ages of 20-44, with a body mass index (BMI) of 20-48, who had a confirmed diagnosis of PCOS from their provider, and exhibited the 2003 Rotterdam criteria for PCOS diagnosis, defined as at least two out of the following three features: clinical or biochemical hyperandrogenism (moderate acne or a modified Ferriman-Gallwey score > 6 or free testosterone > 5 pg/mL), polycystic ovaries (> 12 cysts on one ovary by ultrasound or ovarian volume > 10 mL for one ovary), and menstrual irregularity (defined as < 8 menstrual periods per year or cycles averaging > 35 days in length).

Exclusion Criteria:

* Females who were smokers, had used hormone-based medications within the last 3 months (hormonal contraception, ovulation inducers, anti-androgens) or who were on insulin-sensitizing agents, had another endocrine disorder diagnosis, were pregnant or breastfed within the last 6 months, were diagnosed with a major psychiatric disorder or were on anti-psychotic medication, or who were currently practicing yoga or receiving osteopathic manipulative treatment or acupuncture on a regular basis.

Ages: 20 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change in androgens | After 3 month intervention (immediately after 3 month intervention) compared with pre intervention (initial = 0 months)
  Change in serum androgen levels with intervention

SECONDARY OUTCOMES:
Change in menstrual cycle length | After 3 month intervention (immediately after 3 month intervention) compared with pre intervention (initial = 0 months)
  Change in average time between day 1 of consecutive menstrual cycles after intervention
Change in acne | After 3 month intervention (immediately after 3 month intervention) compared with pre intervention (initial = 0 months)
  Acne score after intervention (none, mild, moderate, severe)
Change in BMI | After 3 month intervention (immediately after 3 month intervention) compared with pre intervention (initial = 0 months)
  BMI value after intervention
Change in waist:hip ratio | After 3 month intervention (immediately after 3 month intervention) compared with pre intervention (initial = 0 months)
  Waist:hip ratio after intervention
Change in fasting blood glucose | After 3 month intervention (immediately after 3 month intervention) compared with pre intervention (initial = 0 months)
  Serum glucose levels after intervention
Change in fasting insulin | After 3 month intervention (immediately after 3 month intervention) compared with pre intervention (initial = 0 months)
  Serum insulin levels after intervention
Change in depression score | After 3 month intervention (immediately after 3 month intervention) compared with pre intervention (initial = 0 months)
  Beck Depression Index II score after intervention (total score 0 to 63, lower score means better outcome)
Change in anxiety | After 3 month intervention (immediately after 3 month intervention) compared with pre intervention (initial = 0 months)
  Beck Anxiety index score after intervention (total score 0 to 63, lower score means better outcome)
Change in blood pressure | After 3 month intervention (immediately after 3 month intervention) compared with pre intervention (initial = 0 months)
  Blood pressure after intervention
Change in heart rate recovery | After 3 month intervention (immediately after 3 month intervention) compared with pre intervention (initial = 0 months)
  Heart rate recovery from exercise after intervention
Change in heart rate variability | After 3 month intervention (immediately after 3 month intervention) compared with pre intervention (initial = 0 months)
  Heart rate variability measured by EKG after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Diana Speelman, Ph.D., Principal Investigator — Lake Erie College of Osteopathic Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Davis SE, Hendryx J, Menezes C, Bouwer S, Menezes H, Patel V, Bostick Smith CA, Speelman DL. Weekly Osteopathic Manipulative Treatment to Improve Measures of Sympathetic Tone in Women With Polycystic Ovary Syndrome: A Randomized, Controlled Pilot Study. J Am Osteopath Assoc. 2020 May 1;120(5):310-321. doi: 10.7556/jaoa.2020.051. PMID 32337566
- [Derived] Patel V, Menezes H, Menezes C, Bouwer S, Bostick-Smith CA, Speelman DL. Regular Mindful Yoga Practice as a Method to Improve Androgen Levels in Women With Polycystic Ovary Syndrome: A Randomized, Controlled Trial. J Am Osteopath Assoc. 2020 Apr 14. doi: 10.7556/jaoa.2020.050. Online ahead of print. PMID 32285088
- [Derived] Davis SE, Hendryx J, Bouwer S, Menezes C, Menezes H, Patel V, Speelman DL. Correlation Between Physiologic and Osteopathic Measures of Sympathetic Activity in Women With Polycystic Ovary Syndrome. J Am Osteopath Assoc. 2019 Jan 1;119(1):7-17. doi: 10.7556/jaoa.2019.004. PMID 30615047